CLINICAL TRIAL: NCT03810755
Title: EfiKroniK Research Program: Effectiveness of Physical Exercise for People With Chronic Pathologies. Hybrid, Clinical and Implementation Randomized Trial
Brief Title: EfiKroniK Research Program: Physical Exercise for People With Chronic Pathologies
Acronym: EfiKroniK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Gonzalo Grandes, Head of the Primary Care Research Unit of Bizkaia, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI17/01172
Record Dates: First submitted 2018-02-26; First posted 2019-01-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Neoplasms; Schizophrenia; COPD; Physical Activity; Quality of Life; Primary Care
MeSH Terms: conditions — Neoplasms; Schizophrenia; Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Experimental: Supervision group= personalized exercise program for patients, supervised during 3 months by nursing in primary and autonomous care afterwards, with support from community resources
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Active Comparator: Control group : PVS program, of proven effectiveness for the promotion of physical activity, diet and smoking cessation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Personalized program (PVS), of proven effectiveness for the promotion of physical activity, diet and smoking cessation.
  Interventions: Other: Personalized Supervised physical activity
- Supervision group (Other): Personalized Supervised physical activity: personalized exercise program for patients, supervised during 3 months by nursing in primary and autonomous care afterwards, with support from community resources
  Interventions: Other: Personalized Supervised physical activity

INTERVENTIONS:
Other: Personalized Supervised physical activity — personalized exercise program for patients, supervised during 3 months by nursing in primary and autonomous care afterwards, with support from community resources

SUMMARY:
Clinical objectives: estimate the common effect of the EfiKroniK physical exercise program for people with a set of Chronic diseases (solid cancers, hematological, schizophrenia and COPD), expressed in terms of functional capacity, quality of life and others results, regarding the standardized intervention of healthy habits 'Prescribe Healthy Living 'PVS.

Implementation objectives: describe the adherence, continuity, adequacy and usefulness of EfiKroniK perceived by patients and professionals, with the purpose of designing implementation strategies, which will be evaluated in future trials.

Design: clinical trial and implementation, pragmatic and randomized to two groups stratified by pathology, followed for 12 m.

Participants: 370 patients diagnosed with solid cancers, hematological cancers, schizophrenia and COPD, in the most advanced stages.

Scope: Hospital de Cruces, Basque Country University, Primary Care Research Unit of Bizkaia.

Intervention: personalized exercise program for patients, supervised during 3 months by nursing in primary and autonomous care afterwards, with support from community resources.

Reference group: PVS program, of proven effectiveness for the promotion of physical activity, diet and smoking cessation.

Measurements: main measure of results: functional capacity at 3 months (6-minute test and submaximal running / running tests at foot to determine the speed of lactate thresholds) and quality of life at 6 and 12 months (SF-36 and specific questionnaires by pathology). Secondary variable results: physical and psychic symptomatology, biological markers, physical form and survival.

Analysis: The common effect of the exercise will be estimated by comparing both groups by intention to treat, by means of analysis of the covariance of mixed effects for the changes observed at 3, 6 and 12 months adjusted for the baseline and possible confounders.

Previously, a possible interaction effect between the pathology group and the effect of the intervention will be ruled out. The cost-effectiveness and cost-utility reasons.

DETAILED DESCRIPTION:
Study design:

This will be a multicentre pragmatic open-label type I hybrid implementation-effectiveness trial, in which a total of 370 patients each with one of 4 different chronic conditions, namely, solid cancer (n=100) and blood cancers (n=70), COPD (n=100) or schizophrenia (n=100), will be randomised to one of two parallel groups, stratified by illness type: the EfiKroniK group (EG) (tailored exercise supervised by fitness and health professionals) or the reference group (PVS group) (36). We deliberately opted to study diverse illnesses seeking to demonstrate any common effect of physical exercise across all of them, independent of any additional effects on each condition separately, and for this purpose, this design is much more efficient than separate clinical trials for each illness. Cardiorespiratory functional capacity at 3, 6 and 12 months and quality of life at baseline at 6 and 12 months will be considered the primary outcome variables, and will compare changes over time in both groups. Additionally, we will explore the perceptions of participants and professionals in terms of the feasibility of the programme, as well as the barriers and facilitators for adherence and continuity.

Study population

Inclusion criteria:

Participants are required to be between 18 and 75 years old and diagnosed with: stage IV solid cancer specifically colon, breast or non-small-cell lung cancer, have an Eastern Cooperative Oncology Group ECOG Performance Status of ≤1, and be on standard first-line chemotherapy; malignant blood cancer and have received an autologous transplant or non-localised lymphoma and be on immune therapy; schizophrenia including first-episode psychosis or other psychotic disorders; or clinically stable (no exacerbation, antibiotic treatment, systemic corticosteroid therapy or hospitalization in the previous 30 days) COPD with a BODE index of 3-7 and a life expectancy >2 years. In addition, the following are required for patients to be eligible for inclusion: good renal, liver and blood function, with haemoglobin levels >10 g/dl, a platelet count > 50,000, neutrophil count > 1,000, and Karnofsky Performance Status score >60, and an Eastern Cooperative Oncology Group Performance Status score ≥ 1.

Exclusion criteria Patients are to be excluded if they have brain metastasis, high risk of fracture due to bone metastasis, severe emotional instability, cardiorespiratory compromise or uncontrolled infection; relapse or progression of blood cancer; alterations in communication or significant cognitive impairment that might hinder data collection; bronchiectasis or lung disease other than COPD; other comorbidities that might hinder or prevent them from following the exercise programme; or uncontrolled high blood pressure (systolic >200 or diastolic >110 mmHg).

Recruitment The Oncology, Haematology and Pulmonology services, primary care doctors and the Mental Health Network of Bizkaia have established an active surveillance system to identify patients with the chronic conditions under study. Doctors will inform patients about the study and invite them to participate. After signing an informed consent form, patients will be referred by the study coordination group to their primary care doctor who will gather baseline data. Before each patient's group allocation is known, a fitness and health professional will measure the study variables at baseline and provide the standardised healthy lifestyle prescription, encouraging physical activity, a balanced diet and smoking cessation.

Randomisation Once informed consent has been obtained and baseline measurements taken, patients will be randomised blindly and centrally to either the EG or PVS group, stratified by illness type, at the coordinating centre, the Primary care Research Unit of Bizkaia of the Biocruces Bizkaia Health Research Institute. The randomization will be performed using computer-generated random numbers in a 1:1 ratio, stratified by illness type, with a block size of 4 or 6.(Fig.1) Protocol for the PVS group On recruitment, all participants will receive a standard healthy lifestyle prescription, encouraging physical activity, a balanced diet and smoking cessation, using the PVS computer tool, which is integrated into the electronic health record. In addition to other measurements at 3, 6 and 12 months, the follow-up will include assessment of potential changes in these habits.

Protocol for the EfiKroniK group First phase: the EfiKroniK group are to participate in an innovative physical exercise programme supervised by fitness and health professionals, ensuring patient safety and adjusting the intensity of the exercise to each patient. In this phase, patients are to develop the skills necessary to become an expert regarding the ideal dose of exercise for them. It consists of 36 sessions of exercise of progressively increasing intensity and tailored to the physical condition of each patient, assessed based on metabolic thresholds. Two sessions a week are to be performed in the laboratory, combining aerobic and strength exercises with stretching, under the supervision of fitness and health professionals and one session a week independently near the health centre, monitored with a HR monitor programmed by the fitness and health professionals. In addition to HR measured with the monitor, exercise is monitored with the modified Borg Rating of Perceived Exertion Scale (37) and the appearance of any symptoms.

Second phase: In this phase, patients are to work independently following a physical exercise programme similar to that of the first phase, taking advantage of resources in the community. To make this feasible, patients are to have been trained during the first phase in the type of exercise and appropriate intensity (Borg Scale,HR monitor, symptoms), and at the end of the 3-month training programme, we will contact individuals who can provide support in the community.

We will calculate the real dose of physical exercise each person has been exposed to: cumulative metabolic equivalent (MET)*h/week and time spent doing moderate and/or vigorous intensity of exercise and intensity of exercise under supervision based on the percentage of heart rate reserve (HRR).

Intensity of aerobic exercise: The American College of Sports Medicine recommends doing at least 150 minutes/week of moderate or 75 minutes/week of vigorous physical activity or a combination of both (38). Regarding the definition of relative intensity, 45-59% of the HRR corresponds to a moderate intensity. Use of this indicator, however, implies carrying out a maximum stress test, the results of which may be distorted by the high degree of fatigue, weakened immune system and reduced peripheral muscle strength of patients who are receiving intensive treatments and have a low level of fitness (28). Furthermore, at the same relative intensity (59% of HRR), the metabolic response varies greatly between individuals (21). For these reasons, we will measure MLs in each patient to allow us to: 1) assess patient aerobic capacity and changes therein, given their strong association with maximum rate of oxygen consumption (VO2max), and 2) ensure patient safety and provide them with a level of metabolic stimulus that is similar across patients and effective in improving biochemical parameters (e.g., reduction in inflammation and improvements in the immune system, blood glucose levels and lipid profile). In particular, the aerobic threshold (LT) can be used in this way given the parallel response between the exponential increase in lactate concentrations that occurs after this LT and the secretion of catecholamines, neurotrophic hormones associated with improvements in cognitive function (BDNF) and anti-inflammatory interleukins (IL-6) involved in reductions in tumour size and reproducibility (39).

The two lactate thresholds will be used as a reference for designing exercise intensity zones for each patient, in terms of speed and HR as well as perceived exertion. The speed at the LT or aerobic threshold determined during an incremental lactate test and the corresponding HR will define the lower limit of the moderate intensity zone. On the other hand, the speed at the threshold, considered the anaerobic threshold, used the measure the maximal lactate steady state (MLSS) (38) and the corresponding HR will be taken as the upper limit of the moderate intensity zone.

Based on the individual MLs, we will design five intensity zones. The zone of low-intensity training (LIT) corresponds to exercise carried out at a HR lower than the LT (~20% of the HRR) and the zone of moderate intensity zone to exercise carried out between the LT and the MLSS (~20-85% of HRR or between 1-2.3 Mmol/L), this in turn being divided into three equally-sized zones: low-moderate (M1), medium-moderate (M2) and high-moderate (M3) intensity. Finally, the zone of high-intensity training (HIT) (>MLSS, >~85% of the HRR).

During the first month, participants will start carrying out sessions involving endurance exercise, which will be divided into 3 intervals of 8 minutes each at an M2 intensity, alternating with 2 minutes at an M1 intensity. In the session in which patients work independently, they will be monitored with HR monitor and it will be explained that they should exercise for 30 minutes and for as much of that time as possible at M1.

During the second month, the maximum intensity of the intervals will increase to M3, nearing the anaerobic threshold HR. Specifically, the fully supervised exercise will be divided into four intervals of 5 minutes at M3, alternating with 3 minutes at M1, while the indirectly monitored (semi-supervised) session will be of 30 minutes at M2 (Figure 2).

Three months after the beginning of the project, the assessments are to be repeated and new intensity zones prescribed, in line with changes in functional capacity as assessed by the lactate tests. At this point, patients are to be given a report of the results of these assessments together with guidelines for exercising independently during the following months. During the same appointment, we will explain to patients how to use the HR zones prescribed during exercise and we will warn them about any potential risk factors detected (39,40). Given that a relatively high proportion of people on the same training programme do not show a good response in various metabolic parameters (41), patients who adapt well to the training will be recommended to continue exercising at a moderate-high intensity (M3), while those with a poorer response will be encouraged to continue their training at least at low- to medium-moderate intensities (M1-M2).

Strength and endurance exercises: Strength training is a key element of the exercise programme in these conditions which are associated with reduced peripheral muscle strength and a low level of fitness. The approach taken consists of exercising the largest muscle groups at high speed and moderate intensity with a moderate load. In each session, 5 exercises are performed involving major muscle groups, namely, the chest, quadriceps, back, hamstring and gluteal muscles, as well as the shoulder, these being performed in 2-3 series of 8-12 repetitions of 16-20 possible exercises (~55-65% of the 1 repetition maximum, seeking to avoid excessive muscle damage and inflammation) and using machines, dumbbells, weight bars and plates, elastic straps and wearable weights.

This type of strength training has shown to be effective for releasing anabolic myokines (IL-4, IL-13, IL-15, leukaemia inhibitory factor) and have great therapeutic potential against osteoporosis and sarcopenia/cachexia (responsible for around 20% of cancer-related deaths) associated with metastatic cancer and associated treatments (39,42), as well as resulting in only mild muscle damage and inflammation.

Outcome measures These measurements are made by an interviewer blind to group allocation.

Primary outcome measure (baseline, 3, 6 and 12 months):

* Cardiorespiratory functional capacity, as assessed using a 400-m walk test
* Changes in health-related quality of life, as assessed using the 36-item Short-Form Health Survey (SF-36) and disease-specific questionnaires: the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) in patients with cancer; and the COPD Assessment Test (CAT) and Chronic Respiratory Disease Questionnaire (CRQ) in patients with COPD.

Secondary outcome measures (baseline, 3, 6 and 12 months):

* Muscle strength test measured by the handgrip strength and sit-and-stand tests
* Thresholds for lactate (LT) and anaerobic threshold or maximal lactate steady state (MLSS), HR, and accelerometer activity counts for tailoring the exercises, determined in submaximal walking or running tests. For detecting the LT, a test will be carried out on a 20-metre track. This will be an incremental test combining 2-minute active period and 1-minute rest period. To help the participant adjust their speed in each 2-minute period, red markers will be placed every 5 metres on the floor and on the wall on both sides and two large cones on the floor at each end of the track. Participants will be asked to reach the next red markers each time they hear a beep, continually adjusting their speed but without stopping; that is, they should go faster or more slowly seeking to pass each set of markers at the time of the corresponding beep. The speed will start at 2.4 km/h in the first stage; and will increase by 0.61 km/h each stage (42). At the end of each stage, the following will be recorded: HR, Rating of Perceived Exertion and lactate concentration, by taking a blood sample from each earlobe to find the minimum lactate equivalent (LEmin) above which the lactate concentration starts to increase exponentially. Hence, the aerobic threshold is defined as the intensity of exercise (speed) at which the lowest recorded lactate level is followed by changes ≥ 0.1 mmol/L in the next stage and >0.2 mmol/L the one after (25). The test will be stopped if the participant becomes exhausted or lactate levels exceed 3 mmol/L.

To identify MLSS, another test will be performed a week after the incremental lactate test to identify the corresponding LT. Based on certain parameters from this progressive test, detailed below, it has been shown to be possible to estimate the speed at which an individual reaches the MLSS accurately (estimates accounting for 86% of the variance in MLSS with standard error of the estimate of 0.385 km/h and the difference between the estimated value of MLSS and the true value lying between -0.77 and 0.81 km/h 95% of the time) (25).

For assessing the MLSS, the patient should return to the health centre where the measurements are taken 1 week later. The infrastructure required is the same as for the incremental lactate test; all that changes is the protocol. An audio recording will be made with two blocks of 10 minutes separated by a 2-minute recovery period, at an MLSS speed estimated using the results obtained in the incremental lactate test and the following equation: MLSS = 3.408 + (1.094·LEmin+1 mM) - (0.036·age - (0.013· LEmin HR)) (25)

* Physical activity performed. For this, each participant will be fitted with an Actigraph wGT3X-BT accelerometer on their right hip at the level of the iliac crest and a HR monitor band (Polar OH1). They should wear these monitors for a week and complete a daily record of their activity, to monitor activity counts during different intensities of activity. To analyse these data, we will assess the activity counts which correlated with the LT during the incremental test and thereby be able to assess their weekly physical activity based on personal activity count thresholds.
* Body composition (OMROM body fat percentage), body mass index and abdominal circumference, estimated cardiovascular risk and the onset of any cardiovascular events
* Psychological changes assessed using Goldberg's 12-item General Health Questionnaire (GHQ-12) and Duke Social Support Index
* In addition, in the case of schizophrenia, changes in mental state assessed using the Positive and Negative Syndrome Scale (PANSS), and the severity of the patient's condition and changes therein during the course of the programme assessed using the Clinical Global Impression (CGI) and the Global Assessment of Functioning (GAF) scale
* Lipid profile, as well as levels of C-reactive protein, glucose, insulin and specific exercise-related parameters: adiponectin, BDNF in participants with schizophrenia, TNF-α in those with cancer and Il-1 and Il-6 in those who have COPD or are transplant recipients (at baseline and 3 months).
* Potential predictive, modifying and confounding factors: sex, age, comorbidities (Adjusted Clinical Groups Case-Mix System), risk factors, socioeconomic status, drug treatments and characteristics of each chronic condition.

ELIGIBILITY:
Inclusion Criteria:

* colon, breast or lung solid cancers stage IV non-small cell, PS ≤1, with standard first-line chemotherapy treatment;
* malignant hemopathy with autologous transplant or lymphomas not localized, in treatment with immunotherapy
* Schizophrenia, including first episodes and other psychotic disorders
* COPD with BODE index 3-7 with clinical stability (absence of exacerbation, antibiotic treatment, systemic corticosteroids or hospitalization, in 30 days prior) and life expectancy> 2 years.
* Adequate renal, hepatic and hematological function, with Hb> 10, platelets> 50,000, neutrophils> 1,000. Karfnosky> 60, ECOG ≥1.

Exclusion Criteria:

* cerebral metastasis
* High risk of fracture due to bone metastasis
* Severe emotional instability
* Cardiorespiratory affectation or uncontrolled infection.
* Relapse or progression of the hematologic disease.
* Altered communication that prevents data collection or important cognitive impairment.
* Bronchiectasis and pulmonary alterations different from COPD.
* Other comorbidities that make it difficult or impossible to carry out the exercise program.
* Unmanaged TA (TAS> 200 or TAD> 110).
* Perform regular physical activity in a intensity, frequency and time equal or superior to the intervention of the supervised program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Functional capacity (6 minute walking test) | One year follow up
  The Test of the 6-minute applies to assess functional capacity, as well as a predictor of morbidity and mortality in people with different pathologies. Most of the daily activities that the patients with these pathologies are performed at submaximal exercise intensity, similar to this test is performed. In addition, as a method of controlling the intensity. Measurements: baseline, at the end of the exercise program, at 6 and 12 months

SECONDARY OUTCOMES:
Change in Health Related Quality of Life: EORTC QLQ- HDC30 in cancer | One year follow up
  The HRQL questionnaire is measured blindly with self-administered questionnaires: EORTC QLQ- HDC30. Measurements: baseline, at the end of the exercise program, at 6 and 12 months
Change in Health Related Quality of Life: CAT and RQ in COPD | One year follow up
  The HRQL questionnaire is measured blindly with self-administered questionnaires: CAT and RQ in COPD. Measurements: baseline, at the end of the exercise program, at 6 and 12 months.
Change in Health Related Quality of Life ( SF36 for all pathologies) | One year follow up
  The HRQL questionnaire is measured blindly with self-administered questionnaires: the Spanish version of the SF-36 and.Measurements: baseline, at the end of the exercise program, at 6 and 12 months.. SF-36 generates an 8-dimension health profile and two summary scores for the physical and mental components. This questionnaire has been validated in the Spanish population.
Change in muscle strength (dynamometer) | One year follow up
  Muscle strength was measured with a handgrip dynamometer adjustable (TKK-5001) in four measurements: baseline, at the end of the exercise program, at 6 and 12 months. The hand grip dynamometry is an objective method for measuring muscle strength and an indicator of the functional integrity of the upper extremity that correlates with overall body strength
Change in biological markers: Concentration of Lipids | 3 months
  Lipids:cholesterol (mg/dl), tryglicerides (mg/dl), HDL (mg/dl), LDL(mg/dl). Measured at baseline, and 3 months
Change in biological markers: Concentration of C reactive protein | 3 months
  C reactive protein (mg/l), Measured at baseline, and 3 months
Change in biological markers: Concentration of glucose | 3 months
  glycemia (mg/dl) Measured at baseline, and 3 months
Change in biological markers: Concentration of Insulin | 3 months
  Insulin (microU/ml). Measured at baseline, and 3 months
Change in biological markers: Concentration of adiponectin | 3 months
  Exercise specific parameters: adiponectin (microgr/mL). Measured at baseline, and 3 months
Change in biological markers: Concentration of BDNF | 3 months
  Exercise specific parameters: BDNF (ng/ml) in mental illness. Measured at baseline, and 3 months
Change in biological markers:Concentration of TNF | 3 months
  Exercise specific parameters: TNF in Cancer patients (pg/ml) .Measured at baseline, and 3 months
Change in biological markers: Concentration of Interleukins II-1 and II-6 | 3 months
  Exercise specific parameters: Interleukins II-1 and II-6 (pg/ml) in COPD patients and transplanted. Measured at baseline, and 3 months
Rates of actate thresholds | One year follow up
  Lactate (mmol/L). Measured at baseline, and 3, 6, 12 months
Change in the physical form | One year follow up
  Measured by an Actigraph xGT3X-BT accelerometer on the right iliac crest and a heart . rate band together with a diary for a week. Measured at baseline, and 3, 6, 12 months
Body composition (fat and muscular weight). (BMI) | One year follow up
  Body Mass Index (BMI): Diagnoses and classifies obesity. weight and height will be combined to report BMI in kg/m^2). Measured at baseline, and 3, 6, 12 months
Psichological changes. Goldberg scale | One year follow up
  It mesures anxiety and Depression. based on responses of 'yes' or 'no' to nine depression and nine anxiety items, asking how respondents have been feeling in the past month. considered patients with anxiety scores of 5 or more or with depression scores of 2 or more as having a 50% chance of a clinically important disturbance. Autoadministered. Measured at baseline, and 3, 6, 12 months
Psichological changes.Duke scale | One year follow up
  To evaluate social suport. It evaluates 2 dimensions: confidential and affective aspects. 11 items, each one with a likert scale (1 to 5 points). Autoadministered. Measured at baseline, and 3, 6, 12 months
Changes in mental health in Schizophrenics. PANSS (Positive and Negative Syndrome Scale) | One year follow up
  PANSS (Positive and Negative Syndrome Scale) .Positive scale: 7 Items, (minimum score = 7, maximum score = 49). Negative scale: 7 items , (minimum score = 7, maximum score = 49). Measured at baseline, and 3, 6, 12 months
Changes in mental health in Schizophrenics. Clinical Gobal Impression (CGI). | One year follow up
  It has 2 scales. 1) Severity scale: 7 ratings ( Normal, not at all ill, Borderline mentally ill, Mildly ill, Moderately ill, Markedly ill, Severely ill, Among the most extremely ill patients). 2) Improvement scale / a 7 point scale). Measured at baseline, and 3, 6, 12 months
Changes in mental health in Schizophrenics. Global activity evaluation (GAF-EEAG) | One year follow up
  A numeric scale to rate subjectively the social, occupational, and psychological functioning of an individual. Scale puntuation: 91 - 100 No symptoms; 81 - 90 Absent or minimal symptoms; 71 - 80 If symptoms are present, they are transient and expectable reactions to psychosocial stressors; 61 - 70 Some mild symptoms; 51 - 60 Moderate symptoms; 41 - 50 Serious symptoms; 31 - 40 Some impairment in reality testing or communication; 21 - 30 Behavior is considerably influenced by delusions or hallucinations or serious impairment; 11 - 20 Some danger of hurting self or others; 1 - 10 Persistent danger of severely hurting self or others; 0 Inadequate information. Measured at baseline, and 3, 6, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Primary care research unit of Bizkaia, Bilbao, Bizkaia, Spain

REFERENCES:
- [Derived] Arietaleanizbeaskoa MS, Sancho A, Olazabal I, Moreno C, Gil E, Garcia-Alvarez A, Mendizabal N, de la Fuente I, Dominguez S, Pablo S, Grandes G; EfiKroniK group. Effectiveness of physical exercise for people with chronic diseases: the EFIKRONIK study protocol for a hybrid, clinical and implementation randomized trial. BMC Fam Pract. 2020 Nov 6;21(1):227. doi: 10.1186/s12875-020-01298-4. PMID 33158422